CLINICAL TRIAL: NCT06457477
Title: The Safety and Efficacy of Sequential Combination Therapy With PD-1 Antibody and Pegylated Interferon-α in NA-supressed Chronic Hepatitis B Patients
Brief Title: Sequential Combination Therapy With PD-1 Antibody and Peg-IFNα in CHB Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIN-CHB-2
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — sintilimab; nas

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody therapy (Experimental)
  Interventions: Drug: Sintilimab; Drug: NAs; Drug: Peg-IFNα-2b

INTERVENTIONS:
Drug: Sintilimab — 100mg/10ml/1bottle
Drug: NAs — tablets
  Other Names: ETV/TDF/TAF
Drug: Peg-IFNα-2b — 180ug/0.5ml/1bottle

SUMMARY:
This is a prospective study to evaluate the safety and efficacy of Sintilimab (PD-1 antibody) in sequential combination with Peg-IFNα-2b in NA-supressed CHB patients who had previously received Peg-IFNα therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 - 65 years old;
* 2.Chronic hepatitis B patients with clear diagnosis of hematology, etiology and clinical (for example: HBsAg positive for more than 6 months);
* 3. In virologically suppressed (HBV DNA below the lower detection limit) CHB patients by NAs treatment, HBsAg decreased by less than 0.5log in the last 6 months of Peg-IFNα therapy, and then discontinued Peg-IFNα at least 6 months;
* 4.Patients with HBV DNA negative, HBeAg negative, HBsAg quantification ≤ 200IU/ml at Peg-IFNα discontinuation and enrollment.

Exclusion Criteria:

* 1. Cirrhosis;
* 2.platelet count < 90×109/L, WBC count < 3.0×109/L, neutrophil count < 1.3×109/L, ALT > ULN (40U/L), total bilirubin > 2ULN;
* 3.History of or suspicion of hepatocellular carcinoma
* 4.Patients received immunosuppressive therapy or other therapy influenced study within 12 months;
* 5.Hepatitis A, hepatitis C, hepatitis D, HIV infection or other active infections;
* 6.Alcohol or drug abuse/dependence;
* 7.Investigator judges that the participants are not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
The rate of HBsAg loss (<0.05 IU/ml) at 24 weeks and 48 weeks | 48 weeks
  Evaluate the level of HBsAg (IU/ml) at 24 weeks and 48 weeks.
Incidence of treatment-emergent adverse events/serious adverse events | 48 weeks
  Evaluate the treatment-emergent adverse events/serious adverse events

SECONDARY OUTCOMES:
The rate of HBsAg decline > 1log(IU/ml) at 24 weeks and 48 weeks | 48 weeks
  Evaluate the level of serum HBsAg (IU/ml) at 24 weeks and 48 weeks.
The rate of HBsAb positive (>10 IU/ml) at 24 weeks and 48 weeks. | 48 weeks
  The rate of HBsAb positive (>10 IU/ml) at 24 weeks and 48 weeks.
The concentration of HBcrAg (logU/mL) at baseline, 12 weeks, 24 weeks and 48 weeks | 48 weeks
  Evaluate the level of serum HBcrAg (logU/mL) at baseline, 12 weeks, 24 weeks and 48 weeks.
The concentration of pgRNA (>10 IU/ml) at baseline, 12 weeks, 24 weeks and 48 weeks | 48 weeks
  Evaluate the level of serum pgRNA (>10 IU/ml) at baseline, 12 weeks, 24 weeks and 48 weeks
The concentration of anti-HBc (IU/ml) at baseline, 12 weeks, 24 weeks and 48 weeks | 48 weeks
  Evaluate the level of serum anti-HBc (IU/ml) at baseline, 12 weeks, 24 weeks and 48 weeks
Immune response of T cell, B cell, NK cell at baseline, 12 weeks, 24 weeks and 48 weeks | 48 weeks
  Evaluate the frequency and function of T cell, B cell, NK cell (tested by flowcytometry/fluorospot/elispot)

CONTACTS AND LOCATIONS:
Locations (1):
- the Fifth Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No